CLINICAL TRIAL: NCT05850156
Title: Study of a Deformability Parameter of Red Blood Cell. FITRED
Brief Title: Study of a Deformability Parameter of Red Blood Cell
Acronym: FITRED
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0433
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Drepanocytosis
MeSH Terms: conditions — Sickle Cell Trait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult sickle cell patients: In the context of routine care, 3 blood collection will be performed on adult sickle cell patients for the analysis of hemoglobin fractions. For each blood collection, an additional volume of blood will be taken for the research purposes.
  Interventions: Procedure: basal blood collection; Procedure: blood collection M6; Procedure: blood collection M12
- pediatric sickle cell patients: In the context of routine care, 3 blood collection will be performed on pediatric sickle cell patients for the analysis of hemoglobin fractions. For each blood collection, an additional volume of blood will be taken for the research purposes.
  Interventions: Procedure: basal blood collection; Procedure: blood collection M6; Procedure: blood collection M12
- Adult sickle cell carriers (heterozygous patients): In the context of neonatal screening for sickle cell disease, the parents will be called altogether with their children in order to check if they are sickle cell carriers or not. Only 1 blood collection will be performed for this group.
  Interventions: Procedure: basal blood collection
- Control patients: In the context of neonatal screening for sickle cell disease, the parents will be called altogether with their children in order to check if they are sickle cell carriers or not. Only 1 blood collection will be performed for this group.
  Interventions: Procedure: basal blood collection

INTERVENTIONS:
Procedure: basal blood collection — blood collection is performed in the context of routine care for hemoglobin analysis. An additional volume of 300µL of blood is taken for the purposes of the study
Procedure: blood collection M6 — 6 months +/- 2 months after inclusion, a blood collection is performed in the context of routine care for hemoglobin analysis. An additional volume of 300µL of blood is taken for the purposes of the study
  Groups: Adult sickle cell patients; pediatric sickle cell patients
Procedure: blood collection M12 — 12 months +/- 2 months after inclusion, a blood collection is performed in the context of routine care for hemoglobin analysis. An additional volume of 300µL of blood is taken for the purposes of the study
  Groups: Adult sickle cell patients; pediatric sickle cell patients

SUMMARY:
Sickle-cell disease is one of the most common severe monogenic disorders in the world, it results in the synthesis of abnormal hemoglobin (HbS) instead of hemoglobin A. When deoxygenated, the sickle haemoglobin (HbS) polymerizes inducing the sickling of red blood cells (RBCs) and leading to decreased deformability and increased fragility. Therefore, sickle RBCs exhibit a reduced lifespan associated with intravascular hemolysis, hemolytic anemia and low tissue oxygenation. Sickle RBCs, which exhibit abnormal adhesive properties to endothelial cells, can block the microcirculation, causing the occurrence of painful vaso-occlusive crisis (VOC), acute chest syndrome (ACS), acute and chronic organ damage (heart, lung, liver, spleen, kidney, bone…) and shortened life span.

A preliminary study performed on RBC from sickle cell patients (Hb SS) has shown an alteration of a parameter measuring the overall deformability of RBCs by evaluating the nature of their movement in a shear flow. This parameter is significantly lower in sickle cell patients in steady state compared to a population of healthy individuals. The parameter is also significantly lower in sickle cell patients during VOC when compared to patient in steady state.

The main objective of this study is to evaluate the performance of the method for measuring the deformability of RBCs on an experimental prototype. Measurements will be performed on blood samples from subjects with a normal hemoglobin electrophoretic profile, from heterozygous carriers of sickle cell disease and from patients with sickle cell disease. Samples from paediatric patients will also be tested to study any specificity in comparison to adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Repeatability of ftt (mechanical marker of deformability) measurements

Exclusion Criteria:

* Effect of ambient temperature on ftt measurements
* Effect of sample processing time on ftt measurements

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric sickle cell patients, adult sickle cell carriers (heterozygous), and adult control subjects (homozygous).
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
repeatability of fTT measurements | 14 months
  A series of 10 measurements of a deformability of red blood cells parameter (fTT) on the same blood sample will be performed successively within 24 hours for 4 samples (2 from sickle cell patient and 2 from control or heterozygous patients). The repeatability of the measurements will be determined from these measurements and the effect of a variation in the total number of red blood cells will be analyzed.This study will be reproduced on several blood samples and the measurements will be repeated under the same conditions 24 hours later.

SECONDARY OUTCOMES:
Effect of ambient temperature during fTT measurement | 14 months
  Tests will be conducted to evaluate the effect of ambient temperature on the measurement of a series of 4 samples at ambient temperature (from 18 to 30°C).
Effect of the processing time on fTT measurement | 14 months
  test will be conducted to measure the fTT on a series of 10 samples, twice a day during the 2 first days an then every day for 5 days.
Correlation of ftt with the collected data | 14 months
  A correlation study of ftt with socio-demographic (age and sex), biological (results of hemogram and hemoglobin electrophoresis) and clinical (number of vaso-occlusive crises and treatment with Hydroxyurea) will be conducted.